CLINICAL TRIAL: NCT00969371
Title: Lenstec TetraFlex Accommodating Posterior Chamber Intraocular Lens (IOL)Clinical Investigation
Brief Title: Lenstec Tetraflex Accommodating Posterior Chamber Intraocular Lens (IOL) Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lenstec Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IDE G050048
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Cataract
Keywords: posterior chamber intraocular lens; PCIOL; IOL
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenstec Tetraflex IOL implantation (Experimental): patients in Study arm received TetraFlex Lens
  Interventions: Device: Experimental TetraFlex Study IOL
- Control IOL (Active Comparator): commercially approved PCIOL implanted
  Interventions: Device: posterior chamber IOL implantation

INTERVENTIONS:
Device: posterior chamber IOL implantation
  Arms: Control IOL
Device: Experimental TetraFlex Study IOL — TetraFlex IOL implanted
  Arms: Lenstec Tetraflex IOL implantation

SUMMARY:
The purpose of the following clinical protocol is to evaluate the safety and effectiveness of the Lenstec Tetraflex Accommodating Posterior Chamber Intraocular Lens (IOL) for the protocol inclusion/exclusion criteria.

DETAILED DESCRIPTION:
The Lenstec TetraFlex Accommodating Posterior Chamber Intraocular Lens (IOL) is an ultraviolet absorbing optical implant designed for the replacement of the human crystalline lens following phacoemulsification cataract removal. The TetraFlex Accommodating Posterior Chamber IOL is designed for treatment of aphakia. The lens is indicated for primary implantation when a cataractous lens has been removed by phacoemulsification with circular tear capsulotomy and the posterior capsule intact. The intended benefit of the TetraFlex Accommodating Posterior Chamber IOL is to provide enhanced distance and near vision with an increased independence from corrective lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Any race
* Patients age at time of surgery to be 18 years or older.
* Presence of bilateral cataract requiring cataract extraction. If only one eye is being implanted with the study lens, the other eye may have had cataract extraction with IOL implantation.
* Clear intraocular media other than cataract.
* Patients with BSCVA < 20/40 or cataract with glare acuity worse than 20/30
* Corneal Astigmatism less than 1 Diopter.
* Good Visual Potential: Best corrected visual acuity (BCVA) projected by PAM or Pinhole 20/25 or better if other pathology is suspected.
* Patient is able and willing to comply with follow-up.
* Able to provide written informed consent.

Exclusion Criteria:

* Patients who are monocular.
* Presence of an ocular infection.
* Greater than or equal to 1 Diopter of pre-operative corneal astigmatism.
* Patients who are on anti-psychotic and antidepressant medication that could potentially effect accommodation
* Patients who chronically take any medication that may affect accommodation, including first generation antihistamines, and anticholinergic agents.
* Previous intraocular surgery in either eye.
* Previous serious corneal disease.
* Diagnosis of any of the following ocular conditions: active scleral disease, glaucoma, retinal disease potentially affecting central vision, macular disease or uveitis, severe dry eyes and dysthyroid eye disease
* Subjects who may be expected to require retinal laser treatment.
* Subjects with diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted to cause future acuity losses to a level of 20/30 or worse).
* Patients requiring administration of topical ophthalmic medications other than the study medications. Use of systemic corticosteroids or anti-metabolites or other medications that could affect wound healing is specifically contraindicated.
* Allergy to anesthetics or other postoperative medications.
* Presence of any uncontrolled systemic disease (e.g. diabetes, hypertension, cardiovascular disease).
* Pregnant or lactating women
* Persons who, in the determination of the investigator, are not competent to understand the procedure, the actions asked of them as research subjects, or capable of completing the patient satisfaction questionnaire.
* Participation in a previous clinical trial within the 30 days prior to the start of the study.
* Persons who may not be able to complete the requirements of returning to the investigator's clinic over the period of the study, or who may be difficult to locate or contact on short notice. This does not preclude vacations or travel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2005-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy outcome is the assessment of the % of eyes obtaining 20/40 or better distance best corrected visual acuity. | 1 year
The primary safety outcome is the incidence/severity of adverse events and complications. | 1 year

SECONDARY OUTCOMES:
Patient's functional reading ability, and other distance, near and intermediate vision testing including subjective patient survey outcomes on dependence on corrective eyewear and patient symptoms. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Sanders, MD, PhD, Study Director — Center for Clinical Research